CLINICAL TRIAL: NCT01223703
Title: Effects of n-3 Polyunsaturated Fatty Acids (PUFAs) on Left Ventricular Function and Functional Capacity in Patients With Dilated Cardiomyopathy
Brief Title: PUFAs and Left Ventricular Function in Heart Failure
Acronym: CS-PUFA-02
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Università degli Studi di Brescia (Other)
Responsible Party: Principal Investigator, Savina Nodari, Effects of n-3 Polyunsaturated Fatty Acids (PUFAs) on Left Ventricular Function and Functional Capacity in Patients With Dilated Cardiomyopathy, Università degli Studi di Brescia
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CS-PUFA-02
Record Dates: First submitted 2010-10-18; First posted 2010-10-19 (Estimated); Results first posted 2011-07-25 (Estimated); Last update posted 2012-01-31 (Estimated); Status verified 2012-01

CONDITIONS: Dilated Cardiomyopathy; Heart Failure
Keywords: n-3 PUFAs; Heart Failure; Dilated cardiomyopathy; Ejection Fraction; Exercise Capacity
MeSH Terms: conditions — Cardiomyopathy, Dilated; Heart Failure | interventions — Omacor

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- n-3 PUFAs (Active Comparator)
  Interventions: Drug: n-3 PUFAs
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: n-3 PUFAs — 1.0 g gelatin capsules containing 850 to 882 mg of EPA and DHA ethyl esters in the average ratio EPA/DHA of 0.9:1.5 The treatment dose was five capsules daily for the first month followed by two capsules daily for the rest of the study.
  Other Names: OMACOR, Pronova Biopharma, Lysaker, Norway
  Arms: n-3 PUFAs
Drug: Placebo — 1.0 g gelatin capsules containing olive oil. The treatment dose was five capsules daily for the first month followed by two capsules daily for the rest of the study
  Arms: Placebo

SUMMARY:
The purpose of this study is to test the hypothesis that n-3 PUFAs improve left ventricular systolic function in patients with stable chronic HF secondary to nonischemic dilated cardiomyopathy (NICM).

DETAILED DESCRIPTION:
The results of the GISSI-HF trial indicate that in patients with chronic HF on evidence-based medical therapy and New York Heart Association (NYHA) functional class II-IV, long term treatment with n-3 PUFAs 1 g daily reduces mortality and hospitalizations for cardiovascular reasons. Several potential mechanisms may underlie the beneficial effects of n-3 polyunsaturated fatty acids (PUFAs) in HF patients, including, but not limited to, antiarrhythmic, and hemodynamic actions. The current investigation was therefore designed to test the hypothesis that treatment with n-3 PUFAs improves LV systolic function expressed as EF in patients with stable chronic HF secondary to a nonischemic dilated cardiomyopathy (NICM). Additionally, we sought to determine if n-3 PUFAs also exert positive effects on LV diastolic function assessed by echocardiography; functional capacity assessed by cardiopulmonary stress testing (CPET); and New York Heart Association (NYHA) functional class.

ELIGIBILITY:
Inclusion Criteria:

* patients with a diagnosis of non ischemic cardiomyopathy (the absence of coronary artery disease,defined as the absence of stenosis > 50%, was confirmed by angiography performed at the time of the diagnostic workup of the cardiomyopathy)
* LV systolic dysfunction (defined as an EF < 45%)
* Stable clinical conditions with minimal or no symptoms for at least three month
* Evidence-based medical treatment at maximum tolerated target doses for at least six month

Exclusion Criteria:

* presence of symptoms or evidence of CAD diagnosed through noninvasive tests;
* peripheral arterial disease;
* presence of congenital or primary valvular heart disease;
* persistent atrial fibrillation;
* inability to perform bicycle ergometry for noncardiac causes;
* moderately to severely reduced functional capacity;
* NYHA functional class IV;
* poor acoustic windows limiting the ability to assess echocardiographic measurements;
* chronic lung disease;
* advanced renal disease (eGFR < 30 mL/min/1.73 m2);
* advanced liver disease;
* any disease limiting life expectancy to one year or less;
* contraindications to study drugs;
* concomitant participation in other research studies

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 133 (Actual)
Dates: Start 2007-11; Primary Completion 2009-06 (Actual); Study Completion 2009-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Savina Nodari, MD, Principal Investigator — Department of Experimental and Applied Medicine-Section of Cardiovascular Diseases; Livio Dei Cas, MD, Study Director — Department of Experimental and Applied Medicine-Section of Cardiovascular Diseases
Locations (1):
- Arrhytmias and Heart failure Unit-Spedali Civili Hospital, Brescia, Italy

REFERENCES:
- [Background] 1.Tavazzi L, Maggioni AP, Marchioli R, et al. Effect of n-3polyunsaturated fatty acids in patients with chronic heart failure (the GISSI-HF trial): a randomised, double-blind, placebo-controlled trial. Lancet2008;372:1223-30. 2.Duda MK, O'Shea KM, Tintinu A, et al. Fish oil, but not flaxseed oil, decreases inflammation and prevents pressure overload-induced cardiac dysfunction. Cardiovasc Res 2009;81:319-27. 3.Duda MK, O'Shea KM, Lei B, et al. Dietary supplementation with omega-3 PUFA increases adiponectin and attenuates ventricular remodeling and dysfunction with pressure overload. Cardiovasc Res 2007;76:303-10. 4.Vargiu R, Littarru GP, Fraschini M, et al. Enhancement of shortening velocity, power, and acto-myosin crossbridge (CB) kinetics following long-term treatment with propionyl-L-carnitine, coenzyme Q10, and omega-3 fatty acids in BIO TO-2 cardiomyopathic Syrian hamsters papillary muscle. Biofactors 2010;36:229-39. 5.Pepe S, McLennan PL. Cardiac membrane fatty acid composition modulates myocardial oxygen consumption and postischemic recovery of contractile function. Circulation 2002;105:2303-8. 6.Duda MK, O'Shea KM, Stanley WC. omega-3 polyunsaturated fatty acid supplementation for the treatment of heart failure: mechanisms and clinical potential. Cardiovasc Res 2009;84:33-41.

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Potential participants were recruited consecutively from the Heart Failure (HF) outpatient clinic of the University of Brescia. The first patient was enrolled on November 5, 2007, and the last patient completed the study on June 30, 2009.
Pre-assignment Details: 458 patients were assessed for eligibility. 235 patients were excluded: 251 not meeting inclusion criteria; 74 refused to participate. A total of 133 patients took part in the study.
Period: Overall Study
Arm/Group | n-3 PUFAs | Placebo
Started | 67 | 66
Completed | 67 | 66
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | n-3 PUFAs | Placebo | Total
Number analyzed (Participants) | 67 | 66 | 133
Age Continuous [Mean (Standard Deviation); unit: years] | 61 (11) | 64 (9) | 62.9 (10.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 10 | 13
  Male | 64 | 56 | 120

OUTCOME MEASURES:

1. Primary Outcome: Change in Left Ventricular (LV) Systolic Function Expressed as Left Ventricular Ejection Fraction (LVEF) Between Baseline and 12-month Follow-up
Description: The primary end point of the study was the change in LV systolic function expressed as LVEF between baseline and 12-month follow-up. The following parameters were measured according to the professional standards defined by the American Society of Echocardiography and the European Association of Echocardiography
Time Frame: one year
Population: A sample of 65 patients in each group was calculated to have 80% power to detect such 0.5 effect size with p<0.05 (2-tailed) at the Student t test for unpaired data.
Measure: Mean (Standard Deviation); unit: ejection fraction (percentage)
Arm/Group | n-3 PUFAs | Placebo
Number analyzed (Participants) | 67 | 66
ejection fraction (percentage)
  baseline | 36 (7) | 37 (6)
  12th month follow up | 39 (6) | 35 (6)
Statistical Analysis 1: Comparison: n-3 PUFAs vs Placebo; null hypothesis is no difference n3 PUFA administration and placebo. To demonstrate an effect size of 0.5 in LVEF, a sample of 65 patients in each group was calculated to have 80% power to detect such 0.5 effect size with alpha=0.05 (2-tailed) at the Student t test. for unpaired data; Test type: Superiority or Other; p < 0.05, t-test, 2 sided; The analysis was done following an intention-to-treat approach by means of the unpaired student t test or Wilcoxon rank sum test as appropriated

2. Secondary Outcome: LV Diastolic Function
Description: Change in LV diastolic function assessed by echocardiography: mitral diastolic inflow velocities (peak velocity of early ventricular filling [E-wave], peak velocity of late ventricular filling [A-wave], E/A ratio, and E-wave deceleration time), diastolic function score (graded on a scale from 1 to 4) were used.
Time Frame: one year
Measure: Mean (Standard Deviation); unit: E/A ratio
Arm/Group | n-3 PUFAs | Placebo
Number analyzed (Participants) | 67 | 66
E/A ratio
  E/A baseline | 0.89 (0.29) | 0.90 (0.37)
  E/A 12 month | 0.84 (0.19) | 0.98 (0.40)
Statistical Analysis 1: Comparison: n-3 PUFAs vs Placebo; Test type: Superiority or Other; p < 0.05, t-test, 2 sided; [statistical method as in outcome 1, analysis 1]

3. Secondary Outcome: Functional Capacity (Change in Peak Oxygen Uptake, VO2)
Description: Change in functional capacity expressed as a peak oxygen uptake (VO2), that was acquired breath-by-breath by pneumotachograph (with bidirectional differential pressure) during cardiopulmonary exercize testing.
Time Frame: one year
Measure: Mean (Standard Deviation); unit: ml/kg/min
Arm/Group | n-3 PUFAs | Placebo
Number analyzed (Participants) | 67 | 66
ml/kg/min
  baseline | 19.5 (3.8) | 18.3 (4.4)
  12th month | 20.7 (4.3) | 17.4 (4.2)

4. Secondary Outcome: Change in Mean New York Heart Association (NYHA) Functional Class Between Baseline and 12th Month Follow up.
Description: NYHA class I: No symptoms and no limitation in ordinary physical activity, e.g. shortness of breath when walking, climbing stairs, etc...
  NYHA class II: Mild symptoms (mild shortness of breath and/or angina) and slight limitation during ordinary activity.
  NYHA class III: Marked limitation in activity due to symptoms, even during less-than-ordinary activity, e.g. walking short distances (20-100 m). Comfortable only at rest NYHA class IV: Severe limitations. Experiences symptoms even while at rest. Mostly bedbound patients.
Time Frame: one year
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | n-3 PUFAs | Placebo
Number analyzed (Participants) | 67 | 66
units on a scale
  baseline | 2.21 (0.51) | 2.17 (0.57)
  12th month | 1.91 (0.54) | 2.32 (0.61)

ADVERSE EVENTS:
Arm/Group | n-3 PUFAs | Placebo
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/67 | 0/66

LIMITATIONS AND CAVEATS:
Our investigation was a single-center trial with a small sample size and a limited number of clinical events. Therefore, our results cannot be generalized to HF patients.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No